CLINICAL TRIAL: NCT00007696
Title: CSP #705D - Screening for Diabetes Mellitus in Veterans
Brief Title: Finding Diabetes Mellitus Among Veterans
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Edelman, David - Study Chair, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: 705D
Record Dates: First submitted 2000-12-29; First posted 2001-01-04 (Estimated); Last update posted 2011-02-03 (Estimated); Status verified 2011-02

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus,DM,glycemic control
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
Population-based screening for diabetes mellitus in non-pregnant adults remains controversial. For a screening strategy to be successful, patients identified by surveillance will have to have better outcomes than if they had been diagnosed at a later, more symptomatic phase of disease. However, little is known about the fate of patients diagnosed with diabetes by screening. Additionally, while about half of the cases of diabetes among the general population at any given time are undiagnosed, the prevalence of undiagnosed diabetes among veterans is unknown. The annual incidence of diabetes among veterans is also unknown.

Assessing risk factors prior to blood testing will improve the specificity, with little cost in sensitivity, of screening for diabetes in a medical center setting. The target population which optimizes the potential value of diabetes screening is patients with at least 1 of the above 3 risk factors for diabetes (obesity, hypertension, family history). Hypertension is strongly associated with unrecognized diabetes in veterans. VA and other health care providers considering whether to perform systematic screening for diabetes should use known risk factors to identify an appropriate target population for screening.

DETAILED DESCRIPTION:
Primary Objectives: To measure the prevalence of undiagnosed Diabetes Mellitus (DM) and the annual incidence of new cases of DM among veterans between the ages of 45 and 64 and to compare the health-related quality of life (HRQoL) of veterans with undiagnosed DM to those without DM but who are at comparable risk for DM, both at baseline and over three years of follow-up.

Secondary Objectives: To describe the clinical state of veterans with diabetes newly diagnosed by screening and to describe the process of usual care for veterans with diabetes newly diagnosed by screening.

Primary Outcomes: The primary outcomes are: 1) prevalence of undiagnosed non-insulin-dependent diabetes mellitus (NIDDM); 2) HRQoL as measured by SF-36; 3) glycemic control as measured by HbA1C; and 4) calculation of the 3-year direct utilization-related cost, from the perspective of the VA, associated with early diagnosis of DM, and comparison of this to the 3-year direct utilization-related cost for veterans who are screened for diabetes but do not have diabetes.

Intervention: N/A

Study Abstract: Population-based screening for diabetes mellitus in non-pregnant adults remains controversial. For a screening strategy to be successful, patients identified by surveillance will have to have better outcomes than if they had been diagnosed at a later, more symptomatic phase of disease. However, little is known about the fate of patients diagnosed with diabetes by screening. Additionally, while about half of the cases of diabetes among the general population at any given time are undiagnosed, the prevalence of undiagnosed diabetes among veterans is unknown. The annual incidence of diabetes among veterans is also unknown.

A mail-out survey for this study was completed with 10,350 surveys mailed and 4,500 surveys returned (43%). Enrollment concluded 7/31/99 with 1,253 new subjects enrolled. Follow-up of the enrolled subjects is ongoing. Some descriptive analyses of the data revealed the prevalence of undiagnosed diabetes was 4.5%. Factors associated with unrecognized diabetes were the diagnosis of hypertension and history of a parent or sibling with diabetes. Having a primary care provider did not raise or lower the risk for unrecognized diabetes. Based on the new diagnosis, most patients found to have diabetes required a change in treatment either of their blood sugar or comorbid hypertension or hyperlipidemia in order to achieve targets recommended in published treatment guidelines. Patients reporting a primary care provider were no less likely to require a change in treatment.

Conclusions: If diabetes screening is an effective intervention, opportunistic screening for diabetes may be the preferred method for screening, as there is substantial potential for case-finding in a medical center outpatient setting. A majority of patients with diabetes diagnosed at opportunistic screening will require a change in treatment of blood sugar, blood pressure, or lipids to receive optimal care.

ELIGIBILITY:
Inclusion Criteria:

Veterans between the ages of 45 and 64.

Exclusion Criteria:

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1276 (Estimated)
Dates: Start 1998-04

CONTACTS AND LOCATIONS:
Overall Officials: David Edelman, MD MHS, Study Chair — Durham VA Medical Center
Locations (1):
- VA Medical Center, Durham, North Carolina, United States